CLINICAL TRIAL: NCT05918809
Title: Real-world Resource Use and Costs of CAR-T Therapies in Diffuse Large B-cell Lymphoma (DLBCL): Inpatient and Outpatient Settings
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019CUS11
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- CAR-T IP: Chimeric antigen receptor modified T cells inpatient cohort
- CAR-T OP: Chimeric antigen receptor modified T cells outpatient cohort
- CAR-T Overall: Chimeric antigen receptor modified T cells overall cohort
- allo-HSCT: Allogeneic hematopoietic stem cell transplant cohort

SUMMARY:
A retrospective, non-interventional cohort study was used to address the study objectives. This study aimed to provide a better understanding of real-world healthcare resource utilization (HRU) and healthcare reimbursement costs associated with chimeric antigen receptor modified T cell (CAR-T) therapy among patients with DLBCL.

ELIGIBILITY:
Inclusion Criteria:

CAR-T cohort:

* Patients had at least one International Classification of Diseases, Tenth Revision (ICD-10) diagnosis code for DLBCL.
* Patients received CAR-T therapy following DLBCL diagnosis. The administration date of CAR-T therapy was defined as the index date. Patients who received both CAR-T therapy and allo-HSCT were classified based on the first treatment that the patient received.
* Patients were at least 18 years of age as of the index date.
* Patients had at least three months of continuous eligibility in the Medicare Part A and Part B data before the index date. Since 2020 Part D data is not available in the current data cut; eligibility requirement in the Part D data was not required.
* Patients were further classified into CAR-T IP and CAR-T OP cohorts depending on where the administration occurred.

Allo-HSCT cohort:

* Patients had at least one ICD-10 diagnosis code for DLBCL.
* Patients received allo-HSCT following DLBCL diagnosis. The date of allo-HSCT procedure was defined as the index date. Patients who received both CAR-T therapy and allo-HSCT were classified based on the first treatment the patient received.
* Patients were at least 18 years of age as of the index date.
* Patients had at least three months of continuous eligibility in the Medicare Part A and Part B data before the index date. Since 2020 Part D data is not available in the current data cut; eligibility requirement in the Part D data was not required.

Exclusion criteria:

• Patients had a medical claim associated with a clinical trial (ICD-9 CM code V70.7; ICD-10 CM code Z00.6) during one month before and after the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1031 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Number of hospital admissions in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Number of inpatient (IP) days in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Number of intensive care unit (ICU) stays in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Number of ICU days in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Number of emergency room (ER) visits in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Number of outpatient (OP) visits in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Percentage of patients in the CAR-T IP and CAR-T OP cohorts with any IP admission | Up to approximately 10 months
Percentage of patients in the CAR-T IP and CAR-T OP cohorts with ER visits | Up to approximately 10 months
Percentage of patients in the CAR-T IP and CAR-T OP cohorts with OP services | Up to approximately 10 months
Total pre-infusion healthcare reimbursement costs in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Total CAR-T infusion-related healthcare reimbursement costs in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months
Total post-infusion healthcare reimbursement costs in the CAR-T IP and CAR-T OP cohorts | Up to approximately 10 months

SECONDARY OUTCOMES:
Cumulative percentage of patients admitted in the hospital during the first month after CAR-T OP infusion | Up to approximately 10 months
Percentage of patients hospitalized each day during the first month after CAR-T infusion among the CAR-T IP and OP cohorts | Up to approximately 10 months
Main cause of IP admission/re-admission among the CAR-T IP and OP cohorts, up to three months following infusion | Up to approximately 10 months
Percentage of patients with AEs | Up to approximately 10 months
Healthcare reimbursement costs per AE event | Up to approximately 10 months
Number of IP admissions in the overall CAR-T and allo-HSCT cohorts | Up to approximately 10 months
Number of IP days in the overall CAR-T and allo-HSCT cohorts | Up to approximately 10 months
Number of OP visits in the overall CAR-T and allo-HSCT cohorts | Up to approximately 10 months
Number of ER visits in the overall CAR-T and allo-HSCT cohorts | Up to approximately 10 months
Total healthcare reimbursement costs in the overall CAR-T and allo-HSCT cohorts | Up to approximately 10 months
Main cause of IP admission/re-admission among the CAR-T IP and OP cohorts | Up to approximately 10 months
Number of intensive care unit (ICU) stays in the overall CAR-T and allo-HSCT cohorts | Up to approximately 10 months
Number of ICU days in the overall CAR-T and allo-HSCT cohorts | Up to approximately 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States